CLINICAL TRIAL: NCT06530901
Title: Multidimensional Ultrasound of the Inferior Vena Cava in the Prevention of Hypotension After Induction of General Anesthesia
Brief Title: Ultrasound of the Inferior Vena Cava in the Prevention of Hypotension After Induction of General Anesthesia
Status: Not yet recruiting | Type: Observational
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Doctor, Yangzhou University
Organization: Yangzhou University (Other)
Other Study IDs: 20240725
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Elderly Patients Undergoing Elective Non-cardiac Surgery
Keywords: hypotension; general anesthesia; inferior vena cava
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients undergoing elective noncardiac surgery under general anesthesia
  Interventions: Diagnostic Test: Multidimensional ultrasound of the inferior vena cava

INTERVENTIONS:
Diagnostic Test: Multidimensional ultrasound of the inferior vena cava — Cross-sectional parameters of the inferior vena cava include two-dimensional longitudinal diameter, cross-sectional length and short diameter, circumference, and cross-sectional area, as well as cross-sectional length and short diameter, circumference, and cross-sectional area in three-dimensional imaging

SUMMARY:
Based on the preoperative ultrasound detection of various parametric indicators of the inferior vena cava cross-section, including the ratio of the inferior vena cava's long and short axes, cross-sectional area and circumference during two-dimensional and three-dimensional imaging, as well as the changes in respiratory variability of each parameter, we explored the predictive value of IVC ultrasound indicator parameters on hypotension after induction of general anesthesia in elderly patients undergoing elective non-cardiac surgery, screened the sensitive indicators, and calculated the cut-off values.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients undergoing elective non-cardiac surgery under general anesthesia;
* Age 65-85 years old;
* Body mass index (BMI) 18-28 kg/m2;
* American society of anesthesiologists (ASA) class I-III.

Exclusion Criteria:

* Patient refusal or lack of cooperation;
* Inability to communicate properly;
* Severe sinus bradycardia, pacemaker implantation, atrioventricular block, and atrial fibrillation;
* Presence of severe hepatic and renal function abnormalities;
* Preoperative cardiac ultrasound suggesting LVEF <50%;
* Tricuspid valve displacement <16 mm by preoperative cardiac ultrasound;
* Chronic obstructive pulmonary disease;
* Pulmonary hypertension;
* Administration of drugs that inhibit the renin-angiotensin-aldosterone system;
* Possibility of a difficult airway.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients undergoing elective non-cardiac surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the level of Mean Arterial Pressure | Baseline (before induction), 10 min after induction
  The outcome above should be measured at the time before induction, 1 min after induction, 2 min after induction, 3 min after induction, 4 min after induction, 5 min after induction,10 min after induction
Changes in the level of Systolic Blood Pressure | Baseline (before induction), 10 min after induction
  The outcome above should be measured at the time before induction, 1 min after induction, 2 min after induction, 3 min after induction, 4 min after induction, 5 min after induction,10 min after induction
Multidimensional ultrasound of the inferior vena cava | Baseline (before induction)
  The outcome above should be measured at the time before induction

SECONDARY OUTCOMES:
Changes in the level of Heart Rate | Baseline (before induction), 10 min after induction
  The outcome above should be measured at the time before induction, 1 min after induction, 2 min after induction, 3 min after induction, 4 min after induction, 5 min after induction,10 min after induction
Changes in the level of Diastolic Blood Pressure | Baseline (before induction), 10 min after induction
  The outcome above should be measured at the time before induction, 1 min after induction, 2 min after induction, 3 min after induction, 4 min after induction, 5 min after induction,10 min after induction

CONTACTS AND LOCATIONS:
Overall Officials: zhuan zhang, professor, Principal Investigator — The Affiliated Hospital of Yangzhou University
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No